CLINICAL TRIAL: NCT01338948
Title: A Feasibility Study on Image-guided Minimally Invasive Robotic Surgery Using Preoperative CT Scan for Gastric Cancer Patients
Brief Title: Image-guided Minimally Invasive Robotic Surgery Using Preoperative CT Scan for Gastric Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: WOO-JIN HYUNG / Associate Professor, Department of Surgery, Yonsei University College of Medicine
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 4-2009-0291
Record Dates: First submitted 2011-03-29; First posted 2011-04-20 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: preoperative 3D-CT reconstruction — Robotic Surgery with CT reconstruction images using Tile-pro program.

SUMMARY:
The purpose of this study is to assess the feasibility of image-guided surgery in patients with early stage gastric cancer using Robotic Surgery with Tile-pro program. For the assessment of the feasibility, conversion to open or laparoscopic surgery due to disturbance of will indicate the failure.

DETAILED DESCRIPTION:
To assess the feasibility of image-guided surgery in patients with early stage gastric cancer using Robotic Surgery with Tile-pro program. For the assessment of the feasibility, conversion to open or laparoscopic surgery due to disturbance of will indicate the failure.

Diagnosis of early stage gastric cancer -> CT scanning & EUS for staging -> (Registration) -> Robotic surgery with image reconstruction -> Conversion rate, Tumor location & vascular anatomy correlation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are older than 20 years
* Histologically confirmed gastric adenocarcinoma
* Patients who want robotic gastric cancer surgery
* Preoperative clinical stage Stage I (T1N0, T1N1, T2N0) diagnosed with EGD, EUS & CT scan
* No history of drug allergy
* creatinine < 1.5 X upper normal limit
* Informed consent

Exclusion Criteria:

* Previous history of upper abdominal surgery
* Patient refused the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
rate of conversion (to laparotomy or laparoscopy assisted) | within 24 hours after operation
  Visualization of upper abdominal vessels (seven vascular structures encountered during gastrectomy)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Matsuki M, Kanazawa S, Kanamoto T, Inada Y, Kani H, Tanikake M, Yoshikawa S, Narabayashi I, Tatsumi Y, Nishimura H, Lee SW, Nomura E, Okuda J, Tanigawa N. Virtual CT gastrectomy by three-dimensional imaging using multidetector-row CT for laparoscopic gastrectomy. Abdom Imaging. 2006 May-Jun;31(3):268-76. doi: 10.1007/s00261-005-0360-2. No abstract available. PMID 16705397
- [Derived] Kim YM, Baek SE, Lim JS, Hyung WJ. Clinical application of image-enhanced minimally invasive robotic surgery for gastric cancer: a prospective observational study. J Gastrointest Surg. 2013 Feb;17(2):304-12. doi: 10.1007/s11605-012-2094-0. Epub 2012 Dec 1. PMID 23207683